CLINICAL TRIAL: NCT04474041
Title: A Clinical Study to Evaluate Visual Acuity Measured With the EyeQue Insight Versus an Eyechart in a Healthcare Office Environment.
Brief Title: Study to Evaluate Visual Acuity Measured With the EyeQue Insight Versus a Standard Eyechart.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeQue Corp. (Industry)
Collaborators: Eye Boutique Optometry (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: EYEQUE - 006
Record Dates: First submitted 2020-07-01; First posted 2020-07-16 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Visual Acuity
Keywords: visual acuity; screening; vision; eye care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Visual Acuity with a Hand-held Device Supported by Mobile App. (Experimental): The Insight will be compared to a standard ETDRS eyechart
  Interventions: Device: EyeQue Insight

INTERVENTIONS:
Device: EyeQue Insight — The Insight will be used to measure visual acuity and compared with a standard ETDRS eye chart.

SUMMARY:
Open label exploratory study of the EyeQue Insight in healthy volunteers >=7 years of age.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether the EyeQue Insight (ETDRS visual acuity test) yields results similar to the standard ETDRS eyechart in the office.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Ages =>7 y.o.
3. Subjects that are minors (<18 years old) must have a parent or legal guardian.
4. Binocular vision
5. Willing and able to give informed consent and follow all study procedures and requirements
6. Fluent in English

Exclusion Criteria:

1. Has been diagnosed within 4 weeks, or currently has signs or symptoms, of COVID-19.
2. Has traveled outside the country within the last 4 weeks
3. Medications:

   a. Taking medications that may affect ability to follow instructions.
4. Eye Disease:

   a. Subjects with eye disease deemed by the Investigator to be inappropriate for the study such as an active eye infection.
5. Subjects that:

   1. Lack physical dexterity to properly operate the EyeQue App on the smartphone
   2. Lack the ability to follow instruction
   3. Lack binocular vision
   4. Lack the ability to maintain both eyes open

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Acuity Visit 1 | Visit 1: Day 0
  Variance of best-corrected (BCVA) monocular VA of each participant's OD and OS measured on the ETDRS chart and the ETDRS test of the EyeQue Insight at Visit 1.

SECONDARY OUTCOMES:
Acuity Visit 1 and 2 | Visit 1 (Day 0) and Visit 2 (Day 7)
  Variance of the best-corrected VA (BCVA) of each participant's OD, OS, and OU measured on the ETDRS chart and the ETDRS test of the EyeQue Insight at Visit 1 and Visit 2.

CONTACTS AND LOCATIONS:
Locations (1):
- EyeQue, Newark, California, United States

IPD SHARING:
Plan to Share IPD: No